CLINICAL TRIAL: NCT01112241
Title: Acute Bronchodilator Responsiveness in Obliterative Bronchiolitis (OB) Following Hematopoietic Stem Cell Transplantation
Brief Title: Bronchodilator Responsiveness in Obliterative Bronchiolitis
Acronym: BD-OB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Responsible Party: Giovanni Barisione, Unit of Preventive and Occupational Medicine - Laboratory of Respiratory Pathophysiology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BOS-01
Record Dates: First submitted 2010-04-27; First posted 2010-04-28 (Estimated); Results first posted 2011-02-23 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2010-04

CONDITIONS: Obliterative Bronchiolitis
Keywords: Obliterative bronchiolitis; Bronchodilator responsiveness; Partial forced expiratory flow; Lung volumes
MeSH Terms: conditions — Bronchiolitis Obliterans | interventions — Albuterol; Tiotropium Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- albuterol-tiotropium (Experimental): At visit 1, lung function measurements will be performed in triplicate before and 90 min after inhaling four separate doses of 100 μg of albuterol (Ventolin®) and soon after 18 μg of tiotropium bromide [Spiriva®] to ensure maximal or near-maximal bronchodilation. Albuterol will be given by a metered-dose inhaler connected to a valved-holding chamber (Volumatic®) and tiotropium by a dry-powder device (Handihaler®).
  Interventions: Drug: albuterol plus tiotropium

INTERVENTIONS:
Drug: albuterol plus tiotropium — Four separate doses of 100 μg of albuterol and 18 μg of tiotropium bromide. Albuterol will be given by a metered-dose inhaler connected to a valved-holding chamber and tiotropium by a dry-powder device.
  Other Names: Ventolin® and Spiriva®

SUMMARY:
This study has been designed to provide a substantial evidence of acute bronchodilator responsiveness to two sequentially inhaled drugs, a beta2-agonist (i.e., albuterol) and an anticholinergic (i.e., tiotropium bromide), in a group of patients who developed obliterative bronchiolitis after hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
Obliterative bronchiolitis is a life-threatening non-infectious pulmonary complication of allogeneic hematopoietic stem cell transplantation (HSCT). It is characterized by the development of an obstructive abnormality which has been considered to be insensitive to bronchodilator treatments. However, this knowledge stems from measurements of forced expiratory volume in 1 s (FEV1) which is relatively insensitive to changes in small airway caliber. Moreover, it is known from studies in chronic obstructive pulmonary disease that symptoms improve after bronchodilator treatment even when FEV1 is minimally increased and correlate with the reduction of lung hyperinflation, which is the major consequence of severe expiratory airflow limitation. Therefore, measurements of airway caliber by parameters not affected by volume history and absolute lung volumes are preferable for assessing the effect of bronchodilator interventions.

In the current study, the bronchodilators responsiveness will be assessed by using not only spirometry but also measurements of absolute lung volumes and the forced expiratory flow of a partial maneuver (V'part) started from submaximal lung inflation, thus free of volume history effects.

ELIGIBILITY:
Inclusion Criteria:

* Obliterative bronchiolitis (OB) following allogeneic HSCT
* FEV1 to slow inspiratory vital capacity (VC) ratio (FEV1/VC)<5th percentile
* FEV1 <75% predicted or absolute FEV1 fall >10% of pre-HSCT value
* evidence of OB by computed tomography scanning
* negative microbiological yields in bronchoalveolar lavage fluid
* chronic graft-versus-host disease score >0
* negative history for bronchial asthma, chronic obstructive pulmonary disease or other significant respiratory disease.

Exclusion Criteria:

* inability to perform lung function maneuvers
* pre-existent chronic lung disease other than OB

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Barisione, MD, Principal Investigator — Unit of Preventive and Occupational Medicine, University Hospital San Martino, Genoa, Italy
Locations (1):
- Unit of Preventive and Occupational Medicine - Laboratory of Respiratory Pathophysiology, University Hospital San Martino, Genoa, Italy

REFERENCES:
- [Background] Pellegrino R, Rodarte JR, Brusasco V. Assessing the reversibility of airway obstruction. Chest. 1998 Dec;114(6):1607-12. doi: 10.1378/chest.114.6.1607. PMID 9872196
- [Background] Barisione G, Bacigalupo A, Crimi E, Van Lint MT, Lamparelli T, Brusasco V. Changes in lung volumes and airway responsiveness following haematopoietic stem cell transplantation. Eur Respir J. 2008 Dec;32(6):1576-82. doi: 10.1183/09031936.0139807. Epub 2008 Aug 6. PMID 18684842
- [Result] Barisione G, Bacigalupo A, Crimi E, Brusasco V. Acute bronchodilator responsiveness in bronchiolitis obliterans syndrome following hematopoietic stem cell transplantation. Chest. 2011 Mar;139(3):633-639. doi: 10.1378/chest.10-1442. Epub 2010 Aug 19. PMID 20724742

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 2010 and May 2010, seventeen consecutive bronchiolitis obliterans (BOS) patients following hematopoietic stem cell transplantation (HSCT) were studied.
Pre-assignment Details: In all patients, airflow obstruction was found at spirometry between 14 and 72 months (median, 41 months) after HSCT. The diagnosis of BOS was confirmed by fulfilment of currently updated criteria [Filipovich AH et al. Biol Blood Marrow Transplant 2005; 11:945-956][Chien JW et al. Biol Blood Marrow Transplant 2010; 16:S106-S114].
Groups:
- Albuterol Plus Tiotropium: At visit 1, lung function measurements will be performed in triplicate before and 90 min after inhaling four separate doses of 100 μg of albuterol (Ventolin®) and soon after 18 μg of tiotropium bromide [Spiriva®] to ensure maximal or near-maximal bronchodilation. Albuterol will be given by a metered-dose inhaler connected to a valved-holding chamber (Volumatic®) and tiotropium by a dry-powder device (Handihaler®).
Period: Overall Study
Arm/Group | Albuterol Plus Tiotropium
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Albuterol Plus Tiotropium
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 48 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Region of Enrollment [Number; unit: participants]
  Italy | 17

OUTCOME MEASURES:

1. Primary Outcome: Per Cent Change of Forced Expiratory Volume in 1 Second (FEV1) After Bronchodilators
Description: Following albuterol plus tiotropium inhalation, FEV1 increments ≥12 per cent as compared to baseline, in an individual subject, were considered as evidence of response to bronchodilators, according to the American Thoracic Society-European Respiratory Society standard criteria [Pellegrino et al. Eur Respir J 2005; 26: 948-968]. They were calculated as follows: [FEV1, expressed in liters (L), after bronchodilators - FEV1 (L) before bronchodilators/FEV1 (L) before bronchodilators x 100].
Time Frame: Baseline and 90 min after bronchodilators
Population: Seventeen consecutive, clinically-stable, Caucasian outpatients, presenting with mild-to-very-severe obliterative bronchiolitis following hematopoietic stem cell transplantation (HSCT) for hematological malignancies, were studied. They were diagnosed from 460 patients (253 males, 207 females) undergoing HSCT (sourcing from bone marrow).
Measure: Mean (Standard Deviation); unit: per cent positive change
Arm/Group | Albuterol Plus Tiotropium
Number analyzed (Participants) | 17
per cent positive change
  Responsives to bronchodilators (n=4) | 14 (1)
  Unresponsives to bronchodilators (n=13) | 7 (5)

2. Primary Outcome: Absolute Change of Forced Expiratory Volume in 1 Second (FEV1) After Bronchodilators
Description: Following albuterol plus tiotropium inhalation, FEV1 increments ≥0.20 liters (L) as compared to baseline, in an individual subject, were considered as evidence of response to bronchodilators, according to the American Thoracic Society-European Respiratory Society standard criteria [Pellegrino et al. Eur Respir J 2005; 26: 948-968]. They were calculated as follows: [FEV1 (L) after bronchodilators - FEV1 (L) before bronchodilators].
Time Frame: Baseline and 90 min after bronchodilators
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: absolute positive change (liters)
Arm/Group | Albuterol Plus Tiotropium
Number analyzed (Participants) | 17
absolute positive change (liters)
  Responsives to bronchodilators (n=4) | 0.26 (0.06)
  Unresponsives to bronchodilators (n=13) | 0.12 (0.09)

3. Primary Outcome: Per Cent Change of Forced Vital Capacity (FVC) After Bronchodilators
Description: Following albuterol plus tiotropium inhalation, FVC increments ≥12 per cent as compared to baseline, in an individual subject, were considered as evidence of response to bronchodilators, according to the American Thoracic Society-European Respiratory Society standard criteria [Pellegrino et al. Eur Respir J 2005; 26: 948-968]. They were calculated as follows: [FVC, expressed in liters (L), after bronchodilators - FVC (L) before bronchodilators/FVC (L) before bronchodilators x 100].
Time Frame: Baseline and 90 min after bronchodilators
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: per cent positive change
Arm/Group | Albuterol Plus Tiotropium
Number analyzed (Participants) | 17
per cent positive change
  Responsives to bronchodilators (n=5) | 24 (13)
  Unresponsives to bronchodilators (n=12) | 2 (4)

4. Primary Outcome: Absolute Change of Forced Vital Capacity (FVC) After Bronchodilators
Description: Following albuterol plus tiotropium inhalation, FVC increments ≥0.20 liters (L) compared with baseline, in an individual subject, were considered as evidence of response to bronchodilators, according to the American Thoracic Society-European Respiratory Society standard criteria [Pellegrino et al. Eur Respir J 2005; 26: 948-968]. They were calculated as follows: [FVC (L) after bronchodilators - FVC (L) before bronchodilators].
Time Frame: Baseline and 90 min after bronchodilators
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: absolute positive change (liters)
Arm/Group | Albuterol Plus Tiotropium
Number analyzed (Participants) | 17
absolute positive change (liters)
  Responsives to bronchodilators (n=5) | 0.65 (0.37)
  Unresponsives to bronchodilators (n=12) | 0.07 (0.15)

5. Primary Outcome: Per Cent Change of Instantaneous Maximal Forced Expiratory Flow (V'Max) After Bronchodilators
Description: Following albuterol plus tiotropium inhalation, V'max increments ≥40 per cent as compared to baseline, in an individual subject, were considered as evidence of response to bronchodilators, according to Pellegrino et al. [Chest 1998; 114:1607-1612]. They were calculated as follows: [V'max, expressed in liters.second-1 (L.s-1), after bronchodilators - V'max (L.s-1) before bronchodilators/V'max (L.s-1) before bronchodilators x 100].
Time Frame: Baseline and 90 min after bronchodilators
Population: Seventeen consecutive, clinically-stable, Caucasian outpatients, presenting with mild-to-very-severe obliterative bronchiolitis following HSCT for hematological malignancies, were studied. They were diagnosed from 460 patients (253 males, 207 females) undergoing HSCT (sourcing from bone marrow).
Measure: Mean (Standard Deviation); unit: per cent positive change
Arm/Group | Albuterol Plus Tiotropium
Number analyzed (Participants) | 17
per cent positive change
  Responsives to bronchodilators (n=4) | 66 (17)
  Unresponsives to bronchodilators (n=13) | 14 (14)

6. Primary Outcome: Per Cent Change of Partial Forced Expiratory Flow (V'Part) After Bronchodilators
Description: Following albuterol plus tiotropium inhalation, V'part increments ≥40 per cent as compared to baseline, in an individual subject, were considered as evidence of response to bronchodilators, according to Pellegrino et al. [Chest 1998; 114:1607-1612]. They were calculated as follows: [V'part, expressed in liters.second-1 (L.s-1), after bronchodilators - V'part (L.s-1) before bronchodilators/V'part (L.s-1) before bronchodilators x 100].
Time Frame: Baseline and 90 min after bronchodilators
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: per cent positive change
Arm/Group | Albuterol Plus Tiotropium
Number analyzed (Participants) | 17
per cent positive change
  Responsives to bronchodilators (n=9) | 59 (26)
  Unresponsives to bronchodilators (n=8) | 17 (7)

7. Primary Outcome: Per Cent Change of Residual Volume (RV) After Bronchodilators
Description: Following albuterol plus tiotropium inhalation, RV decrements ≥10 per cent as compared to baseline, in an individual subject, were considered as evidence of response to bronchodilators, according to O'Donnell et al. [Eur Respir J 2001; 18: 914-920]. They were calculated as follows: [RV, expressed in liters (L), before bronchodilators - RV (L) after bronchodilators/RV (L) after bronchodilators x 100].
Time Frame: Baseline and 90 min after bronchodilators
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: per cent negative change
Arm/Group | Albuterol Plus Tiotropium
Number analyzed (Participants) | 17
per cent negative change
  Responsives to bronchodilators (n=8) | 19 (5)
  Unresponsives to bronchodilators (n=9) | 0 (5)

8. Primary Outcome: Absolute Change of Residual Volume (RV) After Bronchodilators
Description: Following albuterol plus tiotropium inhalation, RV decrements ≥0.30 liters (L) as compared to baseline, in an individual subject, were considered as evidence of response to bronchodilators, according to O'Donnell et al. [Eur Respir J 2001; 18: 914-920]. They were calculated as follows: [RV (L), before bronchodilators - RV (L) after bronchodilators].
Time Frame: Baseline and 90 min after bronchodilators
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: absolute negative change (liters)
Arm/Group | Albuterol Plus Tiotropium
Number analyzed (Participants) | 17
absolute negative change (liters)
  Responsives to bronchodilators (n=8) | 0.65 (0.37)
  Unresponsives to bronchodilators (n=9) | 0.00 (0.10)

9. Primary Outcome: Per Cent Change of Functional Residual Capacity (FRC) After Bronchodilators
Description: Following albuterol plus tiotropium inhalation, FRC decrements ≥10 per cent as compared to baseline, in an individual subject, were considered as evidence of response to bronchodilators, according to O'Donnell et al. [Eur Respir J 2001; 18: 914-920]. They were calculated as follows: [FRC, expressed in liters (L), before bronchodilators - FRC (L) after bronchodilators/FRC (L) after bronchodilators x 100].
Time Frame: Baseline and 90 min after bronchodilators
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: per cent negative change
Arm/Group | Albuterol Plus Tiotropium
Number analyzed (Participants) | 17
per cent negative change
  Responsives to bronchodilators (n=4) | 16 (6)
  Unresponsives to bronchodilators (n=13) | 2 (5)

10. Primary Outcome: Absolute Change of Functional Residual Capacity (FRC) After Bronchodilators
Description: Following albuterol plus tiotropium inhalation, FRC decrements ≥0.30 liters (L) as compared to baseline, in an individual subject, were considered as evidence of response to bronchodilators, according to O'Donnell et al. [Eur Respir J 2001; 18: 914-920]. They were calculated as follows: [FRC (L), before bronchodilators - FRC (L) after bronchodilators].
Time Frame: Baseline and 90 min after bronchodilators
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: absolute negative change (liters)
Arm/Group | Albuterol Plus Tiotropium
Number analyzed (Participants) | 17
absolute negative change (liters)
  Responsives to bronchodilators (n=4) | 0.78 (0.34)
  Unresponsives to bronchodilators (n=13) | 0.07 (0.16)

ADVERSE EVENTS:
Arm/Group | Albuterol Plus Tiotropium
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No